CLINICAL TRIAL: NCT01872286
Title: A Double-center Randomized Head-to-head Comparison of the Frequency-altering AKE-1 Capsule and Pillcam SB2
Brief Title: Comparison of the Frequency-altering AKE-1 Capsule and Pillcam SB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Second Military Medical University (Other); Ministry of Education, China (Other Government)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept., Changhai Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: capsule-1
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Intestinal Diseases; Gastrointestinal Hemorrhage
Keywords: Capsule Endoscopy
MeSH Terms: conditions — Intestinal Diseases; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pillcam SB2 first (Experimental): patients were assigned to swallow PSB first, followed by the AKE
  Interventions: Device: AKE-1; Device: Pillcam SB2
- AKE-1 first (Experimental): patients were assigned to swallow AKE first, followed by the PSB
  Interventions: Device: AKE-1; Device: Pillcam SB2

INTERVENTIONS:
Device: AKE-1
Device: Pillcam SB2

SUMMARY:
Capsule endoscopy has been shown to be the first-line endoscopic procedure for small bowel disease. This study was aimed to compare the performance between the frequency-altering AKE-1 capsule and the Pillcam SB2 in patients with suspected small bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* obscure gastrointestinal bleeding
* chronic diarrhea
* suspected Crohn's disease
* chronic abdominal pain
* neoplastic lesions of small bowel

Exclusion Criteria:

* patients with any contraindication to capsule endoscopy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
judgement of normal or abnormal of gastrointestinal tract | 5 weeks after the examination
  If a lesion is detected by capsule endoscopy in gastrointestinal tract in a patient, the result will be judged as abnormal.

SECONDARY OUTCOMES:
complete small-bowel examination rate | 5 weeks after the examination
diagnostic yield | 5 weeks after the examination
  The finding that could explain the symptom and resulted in clinical impact was considered as diagnosis.Diagnostic yield of a capsule endoscopy is the proportion of patients with positive diagnosis over total patients.
total recording time | 5 weeks after the examination
gastric transit time | the comparison was completed 5 weeks after the examination
small-bowel transit time | the comparison was completed 5 weeks after the examination
total number of images captured | the comparison was completed 5 weeks after the examination

OTHER OUTCOMES:
number of adverse events as a measure of safety | 2 months after the examination

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-Shen Li, Dr., Principal Investigator — Changhai Hospital
Locations (2):
- China (2):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Liao Z, Gao R, Xu C, Li ZS. Indications and detection, completion, and retention rates of small-bowel capsule endoscopy: a systematic review. Gastrointest Endosc. 2010 Feb;71(2):280-6. doi: 10.1016/j.gie.2009.09.031. PMID 20152309
- [Background] Cave DR, Fleischer DE, Leighton JA, Faigel DO, Heigh RI, Sharma VK, Gostout CJ, Rajan E, Mergener K, Foley A, Lee M, Bhattacharya K. A multicenter randomized comparison of the Endocapsule and the Pillcam SB. Gastrointest Endosc. 2008 Sep;68(3):487-94. doi: 10.1016/j.gie.2007.12.037. Epub 2008 Apr 14. PMID 18410941
- [Background] Dolak W, Kulnigg-Dabsch S, Evstatiev R, Gasche C, Trauner M, Puspok A. A randomized head-to-head study of small-bowel imaging comparing MiroCam and EndoCapsule. Endoscopy. 2012 Nov;44(11):1012-20. doi: 10.1055/s-0032-1310158. Epub 2012 Aug 28. PMID 22930176